CLINICAL TRIAL: NCT03131466
Title: Effectiveness and Safety of High-voltage Pulsed Radiofrequency on Gasserian Ganglion to Treat Patients With Primary Trigeminal Neuralgia
Brief Title: High-voltage Pulsed Radiofrequency on Gasserian Ganglion to Treat Patients With Primary Trigeminal Neuralgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Beijing Friendship Hospital (Other); Beijing Ditan Hospital (Other)
Responsible Party: Principal Investigator, Fang Luo, vice director of Department of Anesthesiology and Pain Management, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KY2017-004-01
Record Dates: First submitted 2017-04-22; First posted 2017-04-27 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Idiopathic Trigeminal Neuralgia
Keywords: Trigeminal Neuralgia; Pulsed Radiofrequency; Gasserian Ganglion
MeSH Terms: conditions — Trigeminal Neuralgia | interventions — Nerve Block

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRF Group (Experimental): This group will undergo 42°C high-voltage pulsed radiofrequency treatment.
  Interventions: Device: High-voltage pulsed radiofrequency
- Nerve Block Group (Active Comparator): This group will undergo nerve block treatment with steroid and local anesthesia.
  Interventions: Drug: Nerve block

INTERVENTIONS:
Device: High-voltage pulsed radiofrequency — The manual PRF mode of the pain treatment generator will be turned on, the upper temperature limit will be set at 42°C, the PRF output voltage will be gradually increased to the highest voltage the patient can tolerate, and the patient will be treated for 360 s. After the treatment, 1.4 ml of a mixture of 0.4 mL of normal saline and 1 mL of 1% plain lidocaine will be injected through the needle of the cannula, and before the needle being removed, 0.5 mL of normal saline will be injected.
  Arms: PRF Group
Drug: Nerve block — The radiofrequency generator will be set at the sensory stimulating mode, and the lowest frequency of 0.2 V will be used for 360s-sham PRF treatment, after which 1.4 mL of a mixture of 2 mg of dexamethasone sodium phosphate and 1 mL of 1% plain lidocaine will be slowly injected through the radiofrequency treatment cannula needle. Before the needle being removed, 0.5 mL of normal saline will be injected.
  Arms: Nerve Block Group

SUMMARY:
The study is designed to compare the effectiveness and safety of high-voltage Pulsed radiofrequency and nerve block for the treatment of primary Trigeminal Neuralgia patients with ineffective conservative treatment and explore better non-surgical treatment methods for Trigeminal Neuralgia patients.

DETAILED DESCRIPTION:
Trigeminal neuralgia (TN) is a paroxysmal, lightning-like, severe pain in the facial area innervated by trigeminal nerve. Patients who have failed to achieve benefits from drug treatment could try to undergo nerve block, a traditional conservative treatment. Pulsed radiofrequency (PRF) is a noninvasive pain intervention technique for the treatment of TN. However, its treatment effectiveness has rarely been reported and remains controversial among scholars. A recent single-center preliminary clinical study showed that high-voltage PRF had significant effectiveness in the treatment of TN. However, whether high-voltage PRF treatment can become an optional treatment for TN patients who have failed to achieve benefits from drug treatment still needs to be confirmed with standardized clinical studies by utilizing conservative nerve block treatment as a control. The study is designed to compare the effectiveness and safety of high-voltage PRF and nerve block for the treatment of primary TN patients with ineffective conservative treatment and explore better non-surgical treatment methods for TN patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Primary Trigeminal Neuralgia meets the criteria of the International Classification of Headache Disorders.
* 18-75 years old.
* Response to drug treatment poorly or unable to tolerate the side effects of drugs.
* A BNI pain intensity scale score of IV-V.
* Supposed to undergo neurosurgical intervention according to Trigeminal Neuralgia treatment guidelines.
* Agree to participate in this trial and have signed the informed consent.

Exclusion Criteria:

* Abnormal routine blood, liver or kidney functions, abnormal blood biochemistry test, or coagulation disorders.
* Abnormal electrocardiogram or chest X-ray results.
* Severe cardiopulmonary dysfunction.
* Infection at the puncture site.
* History of mental illness, or history of narcotic drug abuse.
* Allergy to local anesthetic drugs or steroids.
* Cannot cooperate with the treatment.
* History of invasive treatments, such as radiofrequency thermocoagulation, chemical ablation, balloon compression surgery, gamma knife treatment, peripheral denervation or microvascular decompression.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2017-04-28 (Actual); Primary Completion 2020-09-03 (Actual); Study Completion 2021-09-03 (Actual)

PRIMARY OUTCOMES:
Effective rate of Primary Trigeminal Neuralgia treatment | 1 year after operation
  The Barrow Neurological Institute (BNI) pain intensity score will be used to assess pain degree. Pain relief degree will be evaluated as "excellent" (BNI pain score I-II), "good" (BNI pain score III), and "poor" (BNI pain score IV-V). The effective rate=excellent and good pain relief (BNI I - III)/total number of cases * 100%.

SECONDARY OUTCOMES:
Patient satisfaction | 1 day, 1 week, 2 weeks, 1 month, 3 months, 6 months, 1 year and 2 years after operation
  Patient satisfaction score (PSS) score will be used to evaluate patient satisfaction: 0 point indicates unsatisfactory, while 10 points indicates very satisfactory.
Dosage of adjuvant antiepileptic drugs | 1 day, 1 week, 2 weeks, 1 month, 3 months, 6 months, 1 year and 2 years after operation
Data regarding patients with a BNI of IV or V who switch to other treatments | 1 day, 1 week, 2 weeks, 1 month, 3 months, 6 months, 1 year and 2 years after operation
Adverse events | 1 day, 1 week, 2 weeks, 1 month, 3 months, 6 months, 1 year and 2 years after opeartion
  Data regarding intraoperative and postoperative adverse events.
The postoperative response rate | 1 day, 1 week, 2 weeks, 1 month, 3 months, 6 months and 2 years after opeartion
  The Barrow Neurological Institute (BNI) pain intensity score will be used to assess pain degree. Pain relief degree will be evaluated as "excellent" (BNI pain score I-II), "good" (BNI pain score III), and "poor" (BNI pain score IV-V). The effective rate=excellent and good pain relief (BNI I - III)/total number of cases * 100%.

CONTACTS AND LOCATIONS:
Overall Officials: Fang Luo, M.D., Principal Investigator — Beijing Tiantan Hospital
Locations (3):
- China (3):
  - Beijing Ditan Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Beijing, Beijing Municipality
  - Beijing Tiantan Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nader A, Kendall MC, De Oliveria GS, Chen JQ, Vanderby B, Rosenow JM, Bendok BR. Ultrasound-guided trigeminal nerve block via the pterygopalatine fossa: an effective treatment for trigeminal neuralgia and atypical facial pain. Pain Physician. 2013 Sep-Oct;16(5):E537-45. PMID 24077204
- [Background] Nader A, Bendok BR, Prine JJ, Kendall MC. Ultrasound-Guided Pulsed Radiofrequency Application via the Pterygopalatine Fossa: A Practical Approach to Treat Refractory Trigeminal Neuralgia. Pain Physician. 2015 May-Jun;18(3):E411-5. PMID 26000688
- [Background] Elsheikh NA, Amr YM. Calcitonin as an Additive to Local Anesthetic and Steroid Injection Using a Modified Coronoid Approach in Trigeminal Neuralgia. Pain Physician. 2016 Sep-Oct;19(7):457-64. PMID 27676662
- [Background] Tsou HK, Chao SC, Wang CJ, Chen HT, Shen CC, Lee HT, Tsuei YS. Percutaneous pulsed radiofrequency applied to the L-2 dorsal root ganglion for treatment of chronic low-back pain: 3-year experience. J Neurosurg Spine. 2010 Feb;12(2):190-6. doi: 10.3171/2009.9.SPINE08946. PMID 20121355
- [Background] Fang L, Ying S, Tao W, Lan M, Xiaotong Y, Nan J. 3D CT-guided pulsed radiofrequency treatment for trigeminal neuralgia. Pain Pract. 2014 Jan;14(1):16-21. doi: 10.1111/papr.12041. Epub 2013 Feb 21. PMID 23433058
- [Background] Luo F, Meng L, Wang T, Yu X, Shen Y, Ji N. Pulsed radiofrequency treatment for idiopathic trigeminal neuralgia: a retrospective analysis of the causes for ineffective pain relief. Eur J Pain. 2013 Sep;17(8):1189-92. doi: 10.1002/j.1532-2149.2012.00278.x. Epub 2013 Jan 16. PMID 23322665
- [Background] Fang L, Tao W, Jingjing L, Nan J. Comparison of High-voltage- with Standard-voltage Pulsed Radiofrequency of Gasserian Ganglion in the Treatment of Idiopathic Trigeminal Neuralgia. Pain Pract. 2015 Sep;15(7):595-603. doi: 10.1111/papr.12227. Epub 2014 Jun 23. PMID 24954016
- [Background] Maarbjerg S, Di Stefano G, Bendtsen L, Cruccu G. Trigeminal neuralgia - diagnosis and treatment. Cephalalgia. 2017 Jun;37(7):648-657. doi: 10.1177/0333102416687280. Epub 2017 Jan 11. PMID 28076964
- [Derived] Jia Y, Cheng H, Shrestha N, Ren H, Zhao C, Feng K, Luo F. Effectiveness and safety of high-voltage pulsed radiofrequency to treat patients with primary trigeminal neuralgia: a multicenter, randomized, double-blind, controlled study. J Headache Pain. 2023 Jul 18;24(1):91. doi: 10.1186/s10194-023-01629-7. PMID 37464283